CLINICAL TRIAL: NCT07336446
Title: A Phase I/II, Modular, Open-Label, Multi-Centre Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of AZD9750 as Monotherapy and in Combination With Other Anticancer Agents in Participants With Metastatic Prostate Cancer (ANDROMEDA)
Brief Title: A Trial to Learn How Safe AZD9750 is and How Well it Works in People With Metastatic Prostate Cancer When Given With or Without Other Anticancer Drugs
Acronym: ANDROMEDA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7270C00001
Record Dates: First submitted 2025-12-19; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Metastasic Prostate Cancer; Prostate Cancer; Androgen Receptor; Proteolysis-targeting chimeras (PROTACs)
MeSH Terms: conditions — Prostatic Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — AZD5305

STUDY DESIGN:
Intervention Model Description: First-in-human, modular, open-label, Phase I/II study with sequential assignment across modules and parts: Part A (monotherapy dose escalation or combination dose finding) and Part B (dose optimization and expansion), evaluating AZD9750 as monotherapy and in combination with saruparib in participants with metastatic prostate cancer.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Module 1 / Part A1 (Experimental): AZD9750 Monotherapy (Dose Escalation) - No randomization
  Interventions: Drug: AZD9750
- Module 1 / Part A2 (Experimental): AZD9750 Monotherapy (Backfills) - No randomization
  Interventions: Drug: AZD9750
- Module 1 / Part B1 (Experimental): AZD9750 Monotherapy (Dose Optimization) - Randomization
  Interventions: Drug: AZD9750
- Module 1 Part B2 (Experimental): AZD9750 Monotherapy (Dose Expansion) - No randomization
  Interventions: Drug: AZD9750
- Module 1 / Part B3 (Experimental): AZD9750 Monotherapy (Dose Expansion) - No randomization
  Interventions: Drug: AZD9750
- Module 2 / Part A (Experimental): AZD9750 + Saruparib (Combination Dose Finding) - No Randomization
  Interventions: Drug: AZD9750; Drug: AZD5305
- Module 2/ Part B (Experimental): AZD9750 + Saruparib (Combination Dose Expansion) - No Randomization
  Interventions: Drug: AZD9750; Drug: AZD5305

INTERVENTIONS:
Drug: AZD9750 — AR-PROTAC
Drug: AZD5305 — PARP1-selective inhibitor
  Other Names: Saruparib
  Arms: Module 2 / Part A; Module 2/ Part B

SUMMARY:
ANDROMEDA is a first-in-human, Phase I/II, open-label, multicenter study of AZD9750 in participants with metastatic prostate cancer. The trial evaluates safety, tolerability, pharmacokinetics/pharmacodynamics, and preliminary efficacy of AZD9750 as monotherapy and in combination with saruparib.

DETAILED DESCRIPTION:
This first-in-human (FiH), Phase I/II, open-label, multicenter study will evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of AZD9750 as monotherapy and in combination with saruparib in participants with metastatic prostate cancer. Additional combinations with other anticancer agents may be added via protocol amendment as separate modules. The study follows a modular design, allowing initial assessment of safety, tolerability, and preliminary efficacy across multiple treatment arms. Each Module has 2 parts: Part A (monotherapy dose escalation or combination dose finding) and Part B (monotherapy dose optimization and expansion or combination dose expansion). Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study intervention occur.

ELIGIBILITY:
* Inclusion Criteria:

  * Participant must be ≥18 years or the legal age at the time of signing the informed consent form.
  * Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate.
  * Documented metastatic disease.
  * Serum testosterone levels ≤ 50 ng/dL.
  * Evidence of disease progression with one of the following:

    1. PSA progression defined by a minimum of 3 rising PSA levels with an interval of ≥ 1 week between each determination.
    2. Radiographic progression of soft tissue disease by RECIST v1.1 with or without PSA progression.
    3. Radiographic progression of bone metastasis with 2 or more documented new bone lesions on a bone scan with or without PSA progression.
  * ECOG performance status score of 0 or 1.
  * Adequate bone marrow and organ function.
  * Part A (Module 1)

    * (a) Part A1 dose escalation: at least 1 prior ARPI and, if applicable, at least 1 taxane-based chemotherapy (regardless of whether in HSPC or CRPC setting).
    * (b) Part A2 backfill: at least 1 but no more than 2 prior ARPIs and, if applicable, at least 1 but no more than 2 prior taxane-based chemotherapies (regardless of whether in HSPC or CRPC setting).
  * Part B (Module 1)

    * (a) B1/B2 dose optimization/expansion: at least 1 but no more than 2 prior ARPIs and, if applicable, at least 1 but no more than 2 prior taxane-based chemotherapies (regardless of whether in HSPC or CRPC setting).
    * (b) B3 dose expansion (no taxane cohort): at least 1 but no more than 2 prior ARPIs for metastatic prostate cancer (regardless of whether in HSPC or CRPC setting). No prior taxane is allowed for inclusion in this cohort.
* Exclusion Criteria:

  * Participants with pathological finding consistent with any presence of small cell carcinoma, predominant neuroendocrine carcinoma, or any predominant histology other than prostate adenocarcinoma.
  * Brain metastases, or spinal cord compression.
  * Any clinically significant cardiac disorders including QT prolongation, abnormal electrocardiogram (ECG).
  * Any clinically significant cardiovascular diseases including symptomatic heart failure, uncontrolled hypertension, acute coronary syndrome, cardiomyopathy, valvular heart disease, atrial fibrillation, stroke.
  * Active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism of AZD9750 and relevant combination IMPs.
  * Participants with any known predisposition to bleeding (eg, active peptic ulceration, recent [within 6 months] hemorrhagic stroke, proliferative diabetic retinopathy).
  * Prior treatment with an AR-PROTAC.

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, as assigned at birth, inclusive of all gender identities
Enrollment: 300 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2029-01-04 (Estimated); Study Completion 2029-01-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicity (DLT), as defined in the protocol (Part A only) | From first dose of study intervention to 28 days post first dose
  To evaluate the safety and tolerability and determine the MTD and/or the RDE(s)/RP2D of AZD9750 as a monotherapy and in combination with other anticancer agents in participants with mCRPC. A DLT is a toxicity defined by the study protocol that occurs from the first dose of study intervention up to the end of the DLT evaluation period that is assessed as clearly unrelated to the primary disease or intercurrent illness.
Number of participants with Adverse Events and Serious Adverse Events | From first dose of study intervention up to 37 days after the last dose of study treatment
  The number of participants with adverse events and with serious adverse events will be assessed.
Number of participants with Adverse Events leading to discontinuation of study intervention | From first dose of study intervention up to 37 days after the last dose of study treatment
  The number of participants with clinically significant changes from baseline in vital signs will be assessed.
Clinically significant changes from baseline in vital signs. | From first study dose up to 37 days after the last dose of study treatment
  The number of participants with clinically significant changes from baseline in vital signs will be assessed.
Clinically significant changes from baseline in physical examination. | From first dose of study intervention up to 37 days after the last dose of study treatment
  The number of participants with clinically significant changes from baseline in physical examination will be assessed.
Clinically significant changes from baseline in ECOG PS. | From first dose of study intervention up to 37 days after the last dose of study treatment
  The number of participants with clinically significant changes from baseline in ECOG PS will be assessed.
Clinically significant changes from baseline in ECGs. | From first dose of study intervention up to 37 days after the last dose of study treatment
  The number of participants with clinically significant changes from baseline in ECGs will be assessed.
Clinically significant changes from baseline in laboratory parameters. | From first dose of study intervention up to 37 days after the last dose of study treatment
  The number of participants with clinically significant changes from baseline in laboratory parameters will be assessed.
Proportion of participants achieving a ≥50% decrease in PSA from baseline (PSA50) (Part B only) | From first dose of study intervention up to 14 days after the last dose of study treatment
  To evaluate the preliminary antitumour efficacy of AZD9750 as monotherapy and in combination with other anticancer agents in participants with mCRPC.

SECONDARY OUTCOMES:
Proportion of participants achieving a ≥ 50% decrease in PSA from baseline (PSA50) (Part A only) | From first dose of study intervention up to initiation of subsequent anticancer therapy (or radiotherapy on target lesions), PSA progression or 14 days after the last dose of study treatment
  To evaluate the preliminary antitumour efficacy of AZD9750 as monotherapy and in combination with other anticancer agents.
Proportion of participants achieving a ≥ 90% decrease in PSA from baseline (PSA90) | From first dose of study intervention up to initiation of subsequent anticancer therapy (or radiotherapy on target lesions), PSA progression or 14 days after the last dose of study treatment
  To evaluate the preliminary antitumour efficacy of AZD9750 as monotherapy and in combination with other anticancer agents.
Objective response rate (ORR) | From randomisation or first dose of study intervention to initiation of subsequent anticancer treatment (or radiotherapy on target lesions) or progression, assessed up to 60 months
  To evaluate the preliminary antitumour efficacy of AZD9750 as monotherapy and in combination with other anticancer agents. ORR will be assessed according to RECIST v1.1 and PCWG3 criteria (bone) and is defined as the percentage of participants who have a confirmed best overall response of CR or PR or NED (in case the subject has neither TLs nor NTLs at baseline) that occurs prior to the initiation of subsequent anticancer treatment (or radiotherapy on target lesions) and prior to progression.
Duration of response (DoR) | From randomisation or first dose of study intervention to the date of first documented radiological disease progression, assessed up to 60 months
  To evaluate the preliminary antitumour efficacy of AZD9750 as monotherapy and in combination with other anticancer agents. DoR is defined as the time from the date of first documented objective response (which is subsequently confirmed) until the date of first documented radiological disease progression or death (by any cause in the absence of disease progression).
Time to response (TTR) | From randomisation or first dose of study intervention to initiation of subsequent anticancer treatment (or radiotherapy on target lesions) or progression, assessed up to 60 months
  To evaluate the preliminary antitumour efficacy of AZD9750 as monotherapy and in combination with other anticancer agents. TTR is defined as the time from randomisation/first dose until the first documentation of a subsequently confirmed objective response prior to progression and prior to starting any subsequent cancer therapy (or radiotherapy on target lesions).
Radiographic progression-free survival (rPFS) | From randomisation or first dose of study intervention to progression, assessed up to 60 months
  To evaluate the preliminary antitumour efficacy of AZD9750 as monotherapy and in combination with other anticancer agents. rPFS is defined as the time from the date of randomisation or first dose until the date of radiographic progression, as assessed per RECIST v1.1 (soft tissue) and/or PCWG3 criteria (bone) and derived from the raw tumour data or death (by any cause in the absence of progression).
Best percentage change in target lesion size from baseline | From screening (Day -28) to initiation of subsequent anticancer treatment (or radiotherapy on target lesions) or progression, assessed up to 60 months
  To evaluate the preliminary antitumour efficacy of AZD9750 as monotherapy and in combination with other anticancer agents. The best change in tumour size from baseline (i.e. depth of response) is the largest decrease from baseline or the smallest increase from baseline in the absence of a reduction and includes all assessments:
  * up to and including the first visit at which the overall visit response is PD,
  * prior to death in the absence of progression,
  * prior to the start of subsequent anti-cancer therapy (or radiotherapy on target lesions)
  * or up to and including the last evaluable RECIST assessment if the subject has not died, progressed or started subsequent anti-cancer therapy (or radiotherapy on target lesions).
Time to PSA response (TTPSA50, TTPSA90) | From first dose of study intervention up to initiation of subsequent anticancer therapy (or radiotherapy on target lesions), PSA progression or 14 days after the last dose of study treatment
  To evaluate the preliminary antitumour efficacy of AZD9750 as monotherapy and in combination with other anticancer agents. TTPSA is defined as the time from randomisation or first dose date until the date of the first documented PSA50 or PSA90 response (which is subsequently confirmed), respectively.
Cmax of AZD9750 | From date of first dose of study intervention up to 115 days after first dose
  To characterize the PK of AZD9750 as monotherapy and in combination with other anticancer agents.
tmax of AZD9750 | From date of first dose of study intervention up to 115 days after first dose
  To characterize the PK of AZD9750 as monotherapy and in combination with other anticancer agents.
AUC of AZD9750 | From date of first dose of study intervention up to 115 days after first dose
  To characterize the PK of AZD9750 as monotherapy and in combination with other anticancer agents.
Cmax of saruparib (Module 2 only) | From date of first dose of study intervention up to 57 days after first dose
  To characterize the PK of saruparib in combination with AZD9750.
Tmax of saruarib (Module 2 only) | From date of first dose of study intervention up to 57 days after first dose
  To characterize the PK of saruparib in combination with AZD9750.
AUC of saruparib (Module 2 only) | From date of first dose of study intervention up to 57 days after first dose
  To characterize the PK of saruparib in combination with AZD9750.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Research Site, Duarte, California
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Nashville, Tennessee
- Research Site, Melbourne, Australia
- Research Site, Vancouver, British Columbia, Canada
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kashiwa